CLINICAL TRIAL: NCT00002501
Title: PHASE II STUDY OF HIGH-DOSE CYCLOPHOSPHAMIDE PLUS RECOMBINANT HUMAN GRANULOCYTE-COLONY STIMULATING FACTOR (rhG-CSF) IN THE TREATMENT OF FOLLICULAR LOW-GRADE NON-HODGKIN'S LYMPHOMA
Brief Title: Cyclophosphamide and Filgrastim in Treating Patients With Stage IV, Relapsed, or Refractory Low-Grade Follicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9150; CLB-9150; CDR0000077861 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-04-22 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Lymphoma
Keywords: stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Filgrastim; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cyclophosphamide + filgrastim (Experimental): Patients receive cyclophosphamide IV over 90 minutes on day 1 and filgrastim (G-CSF) subcutaneously beginning on day 3 and continuing until blood counts recover. Treatment continues every 2 weeks for 4 courses in the absence of disease progression or stable disease. Patients who achieve complete remission (CR) after completion of course 4 receive 2 additional courses. Patients who achieve partial remission (PR) after completion of course 4 receive 2 additional courses, and those who achieve CR after completion of course 6 receive 2 additional courses. Patients are followed every 2 months for 6 months, every 6 months for 2 years, and then annually thereafter.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of cyclophosphamide and filgrastim in treating patients with stage IV, relapsed, or refractory low-grade follicular non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of high-dose cyclophosphamide and filgrastim (G-CSF) in patients with stage IV, relapsed, or progressive low-grade follicular non-Hodgkin's lymphoma. II. Determine the toxic effects of this regimen in these patients, including those with marrow involvement. III. Determine the rates of complete remission (CR) and partial remission and time to failure in previously treated and untreated patients. IV. Determine the effectiveness of this regimen in eradicating bcl-2 rearrangements, as determined by polymerase chain reaction (PCR), in previously untreated patients. V. Correlate the duration of CR to PCR results in responding patients.

OUTLINE: Patients are stratified according to prior treatment (yes vs no). Patients receive cyclophosphamide IV over 90 minutes on day 1 and filgrastim (G-CSF) subcutaneously beginning on day 3 and continuing until blood counts recover. Treatment continues every 2 weeks for 4 courses in the absence of disease progression or stable disease. Patients who achieve complete remission (CR) after completion of course 4 receive 2 additional courses. Patients who achieve partial remission (PR) after completion of course 4 receive 2 additional courses, and those who achieve CR after completion of course 6 receive 2 additional courses. Patients are followed every 2 months for 6 months, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven low-grade non-Hodgkin's lymphoma of the following subtypes: Follicular, predominantly small cleaved cell Follicular mixed (small cleaved and large cell) Previously treated on Protocol CLB 8691 or previously untreated Previously untreated patients with Stage IV disease (Ann Arbor classification) must meet the following conditions: Documented bone marrow involvement Lymph node biopsy must not show higher grade lymphoma At least 1 additional risk factor as follows: At least 2 extranodal sites Nodes or nodal group at least 5 cm Male Previously treated patients must have progressed or relapsed on Protocol CLB-8691 Recurrence should be documented by biopsy if possible Bidimensionally measurable disease by physical exam, radiograph, CT, or MRI (sonography and barium studies alone not acceptable) Measurable liver disease defined as: Mass greater than 3.5 cm on CT, MRI, or ultrasound OR Histologically documented lymphomatous hepatomegaly more than 5 cm below the costal margin The following disease manifestations are not considered measurable: Ascites or pleural effusion Bony disease (lytic lesions on x-ray should be documented and followed) CNS lesions Bone marrow involvement No lymphomatous involvement (including CNS lymphoma) requiring immediate radiotherapy A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 to physiologic 55 Patients over 55 are eligible only if study chairperson agrees that the patient can tolerate intensive chemotherapy Performance status: Zubrod 0-1 Life expectancy: More than 2 years Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin less than 1.5 times normal Renal: Creatinine less than 1.5 times normal Cardiovascular: LVEF at least 50% No acute changes or arrhythmias on ECG No cardiomegaly on chest x-ray or physical exam No uncontrolled or severe cardiovascular disease, including myocardial infarction within the past 6 months or congestive heart failure (CHF) No active cardiac problems, including compensated CHF or angina Other: HIV negative No other malignancy within the past 5 years except curatively treated basal cell skin cancer or carcinoma in situ of the cervix No active uncontrolled bacterial, viral, or fungal infection No other serious medical illness that would limit survival to less than 2 years No psychiatric condition that would preclude informed consent or compliance No uncontrolled duodenal ulcer Not pregnant Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior interferon only on Protocol CLB-8691 allowed Chemotherapy: Prior oral cyclophosphamide only on Protocol CLB-8691 allowed No concurrent chemotherapy Endocrine therapy: No chronic steroids for other health problems No concurrent steroids for any condition including documented CNS metastases, adrenal failure, or septic shock Nonsteroidal hormonal drugs for nondisease related problems allowed (e.g., insulin for diabetes) Radiotherapy: See Disease Characteristics No prior radiotherapy No concurrent palliative radiotherapy Surgery: At least 2 weeks since prior major surgery Other: No other prior therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 1992-10; Primary Completion 2001-07 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Toxicity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Perri, MD, Study Chair — Veterans Affairs Medical Center - Minneapolis
Locations (15):
- United States (15):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee

REFERENCES:
- [Result] Lichtman SM, Petroni G, Schilsky RL, Johnson JL, Perri RT, Niedzwiecki D, Sklar J, Barcos M, Peterson BA. High dose cyclophosphamide plus recombinant human granulocyte-colony stimulating factor (rhG-CSF) in the treatment of follicular, low grade non-Hodgkin's lymphoma: CALGB 9150. Leuk Lymphoma. 2001 Nov-Dec;42(6):1255-64. doi: 10.3109/10428190109097750. PMID 11911406